CLINICAL TRIAL: NCT04865068
Title: Echocardiographic Standards and Sub-Saharian Africans (SSA) Migrants' in New Aquitaine Region: NEMANA
Brief Title: Echocardiographic Standards and Sub-Saharian Africans (SSA) Migrants' in New Aquitaine Region
Acronym: NEMANA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Limoges (Other)
Collaborators: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 87RI20_0020 /NEMANA
Record Dates: First submitted 2021-04-15; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Diagnosis
Keywords: Echocardiography, Diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- African migrant's population located in la region New Aquitaine. (Experimental): Echocardiography norms will be harvested data on SSA participants located in la region New Aquitaine, France
  Interventions: Diagnostic Test: Echocardiography measures on SSA participants

INTERVENTIONS:
Diagnostic Test: Echocardiography measures on SSA participants — Upon SSA Subject is admitted to the hospital for an echocardiography,
  * Information about this study process,
  * Participants will receive an information note ;
  * Administration of a medical history questionnaire, collection of cardiovascular risk factors, weight toe (all of which are routinely collected before an echocardiographic examination is performed);
  * Performing and recording the echocardiographic examination according to routine protocol
  * delivery of the results according to the usual management;
  * deferred analysis of the recordings on workstation with classification of the data (normal-pathological) according to the different standards

SUMMARY:
Standards Echocardiographic have been defined mainly on caucasian or Asian populations. In the EchoNoRMAL study the criteria for African populations were based solely on data from 198 subjects. This study suggests the presence of different standards depending on the ethnic origin of the subjects. The aims of this study is to describe the proportion of subjects reclassified (normal-pathological) according to the use of echocardiographic norm differences showed in TAHES population (Sub Saharian Africans) with those routinely used

DETAILED DESCRIPTION:
Sub-Saharian Africans populations seem to be more vulnerable in the field of health in general and in cardiovascular pathologies in particular.

* The echocardiographic standards were mainly defined for Caucasian or Asian populations (EchoNoRMAL col. 2014 and 2015). In the EchoNoRMAL study, the criteria for the African populations were based on a reduced workforce (data from 198 subjects).
* This study suggests the presence of different standards depending on the ethnic origin of the subjects. The authors noted that the establishment of references according to the ethnic origin of the subjects is necessary and highlighted the need for additional study for the underrepresented groups, in particular those including subjects of African origin.

The need for different ECG standards in African subjects, was confirmed in a study in the general African population (TAHES), represents 16% of immigrants in 2015 (INSEE According to reports from the health insurance funds, the migrant population,

ELIGIBILITY:
Inclusion Criteria:

- SSA Major Subjects (first generation or from or from first generation parents) admitted to the hospital for an echocardiography

Exclusion Criteria:

* Participation refusal;
* Any acute heart disease (endocarditis, myocarditis, coronary syndrome);
* Valvulopathy justifying an intervention;
* Diseases of overload.
* Any acute heart disease (endocarditis, myocarditis, coronary syndrome);
* Valvulopathy justifying an intervention;
* Diseases of overload.
* Both participant and accompanying person unable to understand the information note written in French and in English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects reclassified (from pathological to normal) according to the echocardiographic standard used (reference standard vs. TAHES standard). | 18 months
  Compare the echocardiography standards previously established in TAHES study to those used routinely managed for the population of SSA migrants in la region New Aquitaine, in order to define pathological subjects

SECONDARY OUTCOMES:
Describe the reasons of reclassification, based on the change of echocardiography standards use for the following criteria: left ventricular hypertrophy, left atrial dilatation, aortic dilatation, ascending, right ventricular dilatation | 18 months
  Identification and analyse the number of subjects requalified from pathological to normal) and identify reasons of the reclassifications after the use of the standards

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lacroix, Professor, Principal Investigator — 0033555056391
Locations (1):
- Explorations fonctionnelles vasculaires et angiologie (Hôpital Dupuytren), Limoges, France